CLINICAL TRIAL: NCT02363140
Title: Magnetic Resonance Imaging to Assess Changes in Meniscus Vascularity
Acronym: MOVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: OR11/9770
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Meniscus Tears
Keywords: Musculoskeletal System
MeSH Terms: interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group One patients in age group 18--20 years, (No Intervention): 1. Patients should be aged 18--20 years or 35--45years
  2. Asymptomatic knee for past 6 months.
  3. Painless flexion-extension movements at knee joint.
- Group Two patients in age group 35-45 years, (Active Comparator): 1. Patients should be aged 18--20 years or 35--45years
  2. Asymptomatic knee for past 6 months.
  3. Painless flexion-extension movements at knee joint.
  Interventions: Other: Will undergo a single MRI assessment with intravenous dye
- Group Three Patients aged 75 (Active Comparator): 1. Patients should be aged 75 or older
  2. Knee X-ray showing no more than Kellgren-Lawrence grade II osteoarthrtis
  3. No clinical suspicion of meniscus tear
  4. Painless flexion-extension movements at knee joint.
  Interventions: Other: Will undergo a single MRI assessment with intravenous dye
- Group Four, any age due to undergo a surgical meniscus repair (Active Comparator): 1. Patients should have presented with clinical signs to suggest meniscus tear indicating potential need for surgical meniscus repair
  Interventions: Other: pre and post surgery MRI scan

INTERVENTIONS:
Other: Will undergo a single MRI assessment with intravenous dye
  Arms: Group Three Patients aged 75; Group Two patients in age group 35-45 years,
Other: pre and post surgery MRI scan
  Arms: Group Four, any age due to undergo a surgical meniscus repair

SUMMARY:
The menisci in the knee joint are important for normal functioning of the knee. Meniscus tears are amongst the commonest of injuries to the knee. The pattern and blood supply of the meniscus tears determines the treatment plan and outcome. The surgeon identifies the blood supply to the meniscus tear area during the arthroscopy(key hole operation) and decides the treatment option ie repair versus partial meniscectomy.

This study aims to identify any changes that occur in the meniscus blood supply. The following are the main aims of the 'MOVE'study-

1. Use of non-invasive methods ie MRImaging to assess meniscus vascularity to preoperatively plan treatment and advice patient on recovery.
2. The study would assess changes in meniscus blood supply depending on age of the patient.
3. The study aims to assess the alteration in meniscus blood supply following an arthroscopic(key hole) meniscal repair operation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Group I,II

1. Patients should be aged 18-20 years or 35-45years
2. Asymptomatic knee for past 6 months.
3. Painless flexion-extension movements at knee joint.

Inclusion criteria for Group III

1. Patients should be aged 75 or older
2. Knee X-ray showing no more than Kellgren-Lawrence grade II osteoarthrtis
3. No clinical suspicion of meniscus tear
4. Painless flexion-extension movements at knee joint.

Inclusion criteria for Group IV

1. Patients should have presented with clinical signs to suggest meniscus tear indicating potential need for surgical meniscus repair.

Exclusion Criteria:

1. Proven Polyarthritis / Polyarthralgia secondary to Rheumatoid arthritis, Gout, Lupus, Ankylosing Spondylosis, Psoriatic arthritis
2. Any previous surgical procedure(open or arthroscopic) involving the knee joint.(baring the current meniscus repair in Group IV participants)
3. Patients unable to give informed consent.
4. Patients with contraindication for MR Imaging - Metal implants, prosthetic heart valves, pacemakers, metal foreign bodies, VP shunts, pregnancy, cochlear implant, metal clips in the brain, Patients with static tremor i.e. Parkinson's disease.
5. Patients with contraindications for contrast agent - Renal impairment, Previous allergic reaction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome is to assess meniscus vascularity in-vivo by use of MR imaging technique. | 6 months